CLINICAL TRIAL: NCT07117461
Title: A Pilot Distress Screening and Referral Program to Detect Comorbid Psychosocial Distress in NYC Safety Net Hospitals Serving Diverse and Underserved Patients Diagnosed With Cancer
Brief Title: A Study of a Distress Screening and Referral Program in People With Recently Diagnosed Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-296
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor Cancer
Keywords: Solid Tumor Cancer; 24-296; Memorial Sloan Kettering Cancer Center

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with a New Solid Tumor Diagnosis (Experimental): Participants will have a new solid tumor cancer diagnosis.
  Interventions: Behavioral: NCCN Distress Thermometer

INTERVENTIONS:
Behavioral: NCCN Distress Thermometer — A tool used to determine on a number scale the amount of distress for the past week

SUMMARY:
It is recommended that cancer centers screen patients for distress and refer them to mental health services when their distress levels reach a certain level. However, many cancer centers don't have distress screening and referral programs. This study will provide valuable information about one distress screening and referral program and whether it can be helpful for a large and diverse group of cancer patients that includes both English- and Spanish-speaking patients.

ELIGIBILITY:
Inclusion Criteria:

* New solid tumor cancer diagnosis (per EMR)
* Treated or will be treated at Jamaica Hospital Medical Center (per EMR)
* Has a NCCN DT score of 0 through 10 (per EMR)
* Age ≥ 18 years (per EMR or self-report)
* English- or Spanish preferred language for healthcare (per self-report)
* Able to provide consent (per completion of consent)

Exclusion Criteria:

* In the provider or investigative teams' judgement, cognitively not intact to participate in the study (per EMR or investigative team)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
Participant referral rate to mental health services | 3 months
  To track outcomes of a pilot distress screening and referral program at Jamaica Hospital Medical Center with English- and Spanish-speaking cancer patients (n=50), by assessing referral rate to mental health services.

CONTACTS AND LOCATIONS:
Overall Officials: Devika Jutagir, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Medisys Health Network (Data Collection Only), Richmond Hill, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org